CLINICAL TRIAL: NCT00588393
Title: Study of the Efficacy and Safety of FolateScan (Technetium TC99m EC20) in Patients With Rheumatoid Arthritis and Other Inflammatory Diseases
Brief Title: FolateScan in Autoimmune Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Endocyte (Industry)
Responsible Party: Eric L. Matteson, M.D., M.P. H., Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 06-002680
Record Dates: First submitted 2007-12-22; First posted 2008-01-08 (Estimated); Last update posted 2010-04-16 (Estimated); Status verified 2010-04

CONDITIONS: Rheumatoid Arthritis; Osteoarthritis; Multiple Sclerosis; Crohn's Disease; Systemic Lupus Erythematosus
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis; Multiple Sclerosis; Crohn Disease; Lupus Erythematosus, Systemic

INTERVENTIONS:
Drug: FolateScan (Technetium Tc 99mEC20) — 0.1 mg. of EC20 labeled with 20-25 mCi of technetium-99m followed by FolateScan

SUMMARY:
This study will gather information on the safety of FolateScan and the ability of FolateScan to detect inflammation in the joints and other organs in people with arthritis (rheumatoid arthritis and osteoarthritis), systemic lupus erythematosus, multiple sclerosis, interstitial pneumonitis, Crohn's disease as well as in healthy persons without these conditions.

DETAILED DESCRIPTION:
The folate receptor is over-expressed on many types of cancer cells and in RA models, and new folate receptor targeted therapies are being developed to target cancer cells that over-express the folate receptor. As with other targeted therapies, it is important to develop diagnostic tests that will provide accurate information on folate receptor status and aid in selecting patients that may benefit from folate-targeted therapy.

EC20 concentrates in the extremities and liver and spleen of rats with adjuvant induced arthritis. The increased uptake is mediated by overexpressed folate receptor on macrophages, and the intensity of the uptake is greatly reduced by addition of excess folate, supporting the specificity of the uptake. Depletion of macrophages greatly reduced folate receptor and abolishes uptake of EC20. This suggests that EC20 may be useful in assessing macrophage involvement in the active inflammatory process of RA, and perhaps other systemic immune mediated disorders as well.

FolateScan may allow the clinician to get accurate real-time data on receptor binding, in a less invasive manner, at all actively inflamed sites throughout the treatment regimen. This kind of information may help the physician make better clinical decisions regarding therapy, including folate targeted therapies.

ELIGIBILITY:
Inclusion Criteria:

* Study will include 40 subjects with rheumatoid arthritis (active or inactive disease, defined as no swollen joints) and 5 patients in each of the following diagnosis: osteoarthritis, multiple sclerosis, Crohn's disease, systemic lupus erythematosus, interstitial lung disease and no autoimmune disease (healthy).
* Subjects must have disease duration of at least 6 months and creatinine level may not be greater than 1.5 mg/dL.

Exclusion Criteria:

* Subjects will be excluded if they are pregnant, have an active infection, received an investigational therapy in the past month or previous malignancy within the past 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2006-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
detection of joint inflammation due to active rheumatoid arthritis | 1 hour post injection of 0.1 mg of EC20

SECONDARY OUTCOMES:
detection of systemic organ inflammation due to rheumatoid arthritis | 1 hour post injection of 0.1mg of EC20

CONTACTS AND LOCATIONS:
Overall Officials: Eric L Matteson, M.D., M.P.H., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Xia W, Hilgenbrink AR, Matteson EL, Lockwood MB, Cheng JX, Low PS. A functional folate receptor is induced during macrophage activation and can be used to target drugs to activated macrophages. Blood. 2009 Jan 8;113(2):438-46. doi: 10.1182/blood-2008-04-150789. Epub 2008 Oct 24. PMID 18952896